CLINICAL TRIAL: NCT07317505
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of JMT108 Injection in Participants With Advanced Malignant Tumors
Brief Title: A Phase 1 Study of JMT108 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JMT108-002
Record Dates: First submitted 2025-11-25; First posted 2026-01-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Cancer (Solid Tumors)
Keywords: cancer; solid tumors; advanced malignant; colorectal cancer; hepatocellular cancer; gastric cancer; melanoma
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Liver Neoplasms; Stomach Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a Dose Escalation (Experimental): In the dose escalation phase, dose escalation will be conducted using a BOIN design. A total of 4 dose levels-0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, and 2 mg/kg-will be sequentially escalated.
  Interventions: Drug: JMT108
- Phase 1a Dose Expansion (Experimental): During the dose escalation process, dose expansion and/or exploration of different dosing frequencies (e.g., Q3W) will be conducted for the dose level that the SMC evaluates as safe/ tolerable and where anti-tumor activity is also observed.
  Interventions: Drug: JMT108
- Phase 1b Cohort Expansion (Experimental): Participants may be enrolled in the cohort expansion study with tumor types including but not limited to Cohort 1: lung cancer, Cohort 2: colorectal cancer, Cohort 3: hepatic cancer, Cohort 4: gastric cancer, Cohort 5: melanoma and Cohort 6: other malignant tumors (including cervical cancer, renal cancer, bile duct cancer, squamous cell head and neck cell cancer, etc.). Based on the results of Phase 1a, the SMC will discuss and determine the administration dose and frequency for the cohort expansion study. If necessary, several different doses/frequencies may be selected for cohort expansion.
  Interventions: Drug: JMT108

INTERVENTIONS:
Drug: JMT108 — Administered by intravenous injection

SUMMARY:
The goal of this clinical trial is to test JMT108, a type of drug called a bispecific antibody in adult patients with locally advanced or metastatic solid tumors.

The main questions it aims to answer are:

* To assess the safety and tolerability of JMT108 at increasing doses and determine the dose and schedule to be used in the second part of the study (Phase 1a)
* To assess effectiveness of JMT108 in participants with locally advanced or metastatic tumors (Phase 1b)
* To evaluate how quickly JMT108 is metabolized by the body (pharmacokinetics or PK)
* To evaluate if antibodies to the study drug develop (immunogenicity)
* To evaluate preliminary efficacy to the drug
* To explore the pharmacodynamic (PD) characteristics of JMT108
* To explore the correlation between biomarker levels and preliminary efficacy

Participants will:

* Provide written informed consent
* Undergo screening tests to ensure they are eligible for study treatment
* Attend all required study visits and receive JMT108 by intravenous injection every 2 weeks until the study doctor determines study treatment should be stopped, based on how well a participant is doing on treatment
* Be followed for progression every 3 months for up to 2 years

DETAILED DESCRIPTION:
This Phase 1 study is a single agent, 2-part (including dose escalating and expansion) study conducted in patients with locally advanced or metastatic solid tumors who are unresponsive or intolerant to all standard of care or have no standard of care available.

Dose escalation (Phase 1a) - Dose escalation will be conducted using a BOIN design.

In the dose-escalation phase, a total of 4 dose levels-0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, and 2 mg/kg-will be sequentially escalated. The BOIN design is adopted for the dose-escalation part of this study to determine the MTD. The target toxicity rate for the MTD is 0.3, and the maximum sample size for the dose-escalation BOIN design is 30 participants. Participants are enrolled to receive treatment in cohorts of size 3. Dose escalation and de-escalation decisions are made based on the occurrence of DLTs within the DLT observation window.

After thorough evaluation by the SMC, one or more dose levels may be added between the highest escalated dose level and the next lower dose level for better DLT assessment.

The dose escalation phase includes a screening period (D-28 to D-1), a treatment period, an end of treatment (EOT) visit, and a follow-up period.

Cohort expansion (Phase 1b) - Based on the results of Phase 1a, the administration dose and frequency for the cohort expansion phase of study will be determined. If necessary, several different doses/frequencies may be selected for cohort expansion. Participants may be enrolled in the cohort expansion study with tumor types including but not limited to Cohort 1: lung cancer, Cohort 2: colorectal cancer, Cohort 3: liver cancer, Cohort 4: gastric cancer, Cohort 5: melanoma and Cohort 6: other advanced solid tumors (including cervical cancer, renal cancer, bile duct cancer, head and neck squamous cell head and neck cancer, etc.).

ELIGIBILITY:
Major Inclusion Criteria:

* Age ≥18 years
* Participants with histologically or cytologically confirmed locally advanced or metastatic solid tumors who are unresponsive or intolerant to all standard of care or have no standard of care available
* At least one evaluable tumor lesion according to RECIST v1.1.
* ECOG performance status score ≤2.
* Expected survival ≥ 3 months

Major Exclusion Criteria:

* Active central nervous system metastases and/or leptomeningeal metastases
* AEs from prior therapy which have not recovered to Grade ≤1 or baseline as per NCI CTCAE v5.0

Prior therapy

* Any other unapproved investigational drugs or treatments within 4 weeks prior to the first dose of the investigational drug (C1D1).
* Chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, or other anti-tumor therapies within 4 weeks prior to the first dose of the investigational drug, except in the following situations:

  1. Nitrosoureas or mitomycin C within 6 weeks prior to the first dose of the investigational drug;
  2. Use of oral fluoropyrimidines and small-molecule targeted drugs within 2 weeks or 5 half-lives of the drug (whichever is longer) prior to the first dose of the investigational drug;
  3. Use of herbal medicine/products with anti-tumor indications within 2 weeks prior to the first dose of the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities as assessed by NCI CTCAE v5.0 (excluding cytokine release syndrome, CRS). | through study completion, an average of 1 year
  To evaluate the safety and tolerability of JMT108 to determine the dose and schedule to be used in phase 1b.
Number of participants with Tumor Response as assessed by RECIST version 1.1 criteria | through study completion, an average of 1 year
  To evaluate preliminary efficacy of JMT108 injection as monotherapy in participants with advanced malignant tumors.

SECONDARY OUTCOMES:
JMT108 Pharmacokinetics: Area under the concentration time curve over the dosing interval | through study completion, an average of 1 year
  JMT 108 Pharmacokinetics: Area under the concentration time curve over the dosing interval.
JMT108 Pharmacokinetics: Elimination half-life (t1/2) | through study completion, an average of 1 year
  JMT108 Pharmacokinetics: Elimination half-life (t1/2)
JMT 108 Pharmacokinetics: Clearance (CL) | through study completion, an average of 1 year
  JMT108 Pharmacokinetics: Clearance (CL)
JMT108 Objective response rate (ORR) | through study completion, an average of 1 year
  ORR is defined as the proportion of patients in whom a complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 is observed as best overall response
JMT108 Immunogenicity: Number of participants with anti-drug-antibody (ADA) | through study completion, an average of 1 year
  JMT108 Immunogenicity: Number of participants with anti-drug-antibody (ADA)

OTHER OUTCOMES:
JMT 108 Pharmacodynamics: Changes in immune cell levels: CD8+ T cells, CD4+ T cells, NK cells, PD-1+ immune cells | through study completion, an average of 1 year
  JMT 108 Pharmacodynamics: Changes in immune cell levels: CD8+ T cells, CD4+ T cells, NK cells, PD-1+ immune cells to explore the PD characteristics of JMT108 Injection
JMT 108 Pharmacodynamics: Changes in cytokine levels (including but not limited to): IL-6, IL-8, TNF-α, IFN-γ | through study completion, an average of 1 year
  Changes in cytokine levels (including but not limited to): IL-6, IL-8, TNF-α, IFN-γ to explore the PD characteristics of JMT108 Injection
JMT108 Correlatives: Correlation of baseline PD-L1 expression with anti-tumor activity | through study completion, an average of 1 year
  Correlation of baseline PD-L1 expression with anti-tumor activity to explore the correlation between biomarker levels and preliminary efficacy

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - NEXT Dallas, Dallas, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No